CLINICAL TRIAL: NCT03993977
Title: ROTEM-guided Transfusion Protocol Versus Standard Care in Attempt to Reduce Blood Transfusions in Potentially Curative Major Abdominal and Urological Oncological Surgery
Brief Title: ROTEM-guided Transfusion Protocol in Attempt to Reduce Blood Transfusions in Major Oncological Surgery
Acronym: ROTEM-SUR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to changes in the surgical technique, no potential subjects anymore
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETL R17025
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Blood Loss, Surgical; Blood Loss Requiring Transfusion; Coagulation Defect; Acquired
Keywords: ROTEM; thromboelastometry; blood transfusion; cancer; surgery; abdominal; oncological
MeSH Terms: conditions — Blood Loss, Surgical; Hemostatic Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: 60 patients having a potentially curative abdomino-oncological surgery and reaching an active blood loss of more than 1500 ml are randomized into two groups. One will be treated conventionally, ie. using MTP if necessary, clinical judgement and conventional coagulation tests, the other treated using a ROTEM-based algorithm. Randomization (ratio 1:1 in blocks of 10) between the two groups will be done beforehand. Each paper containing the treatment protocol in question will be put into a closed envelope. The envelopes are numbered from 1 to 60 and are placed in a box in the operative department.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not know which group he/she is randomized into. They are under general anaesthesia, thus not knowing which protocol is used. When assessing outcomes, two groups are labeled only by number: the assessor does not know which arm is number 1 or 2 until whole data is analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROTEM-arm (Experimental): Treatment of significant blood loss using point-of-care testing of whole blood viscoelasticity (ROTEM) monitoring coagulopathy or hyperfibrinolysis.
  Interventions: Diagnostic Test: Rotational thromboelastometry
- Control-arm (Active Comparator): Treatment of significant blood loss conventionally, ie. using massive transfusion protocol if necessary, clinical judgement and conventional coagulation tests, such as prothrombin time (as international normalized ratio, INR), activated partial thrombin time (APTT), fibrinogen in plasma (Clauss method).
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Diagnostic Test: Rotational thromboelastometry — ROTEM-guided protocol of hemostatic resuscitation
  Other Names: ROTEM
  Arms: ROTEM-arm
Other: Conventional treatment — Clinical judgement and conventional coagulation tests
  Arms: Control-arm

SUMMARY:
Need for perioperative blood transfusion is still high in certain types of oncological abdominal surgery. Allogeneic blood transfusion may be detrimental in cancer patients undergoing a potentially curative resection of malignant tumor, although the detailed mechanism of this effect is still under debate. We plan to evaluate whether a new, rotational thromboelastography-guided algorithm (ROTEM) to guide hemostatic resuscitation intra-operatively decreases the use of allogeneic blood products, the total amount of bleeding, transfusion related side effects, thromboembolic complications and costs. Its effect on each patient's post-operative hemostatic profile is also measured. 60 patients having a potentially curative pancreaticoduodenectomy (or resection of cauda of pancreas), total removal or partial resection of kidney and open radical cystectomy are recruited when an active blood loss of more than 1500 ml is estimated and/or measured and are randomized into two groups: one will be treated conventionally, ie. using massive transfusion protocol (MTP) if necessary, clinical judgement and conventional coagulation tests, the other treated using a ROTEM-based algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18, radical cystectomy, total or partial nephrectomy for malignant disease or pancreaticoduodenectomy planned and estimated intraoperative hemorrhage over 1500ml, written and informed consent

Exclusion Criteria:

* Known hemophilia or von Willebrandt's disease (treatment planned beforehand in collaboration with haematologist), unacceptance of allogeneic blood products (jehovah's witnesses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Number of transfused red blood cell (RBC) units | 24 hours after beginning of surgery
  Red blood cell units transfused per patient during operation or up to 24 hours after beginning of surgery

SECONDARY OUTCOMES:
Intensive care admissions | 30 days after surgery
  Number of patients admitted to intensive care or high dependency, if this is considered associating with the surgery
Length of hospital stay | 30 days after surgery
  Number of days patient is in hospital immediately after surgery
Transfusion-related side effects | 30 days after surgery
  Any side-effect considered or suspected originating from blood product transfusion
Thromboembolic events | 30 days after surgery
  Clinically diagnosed deep vein thrombosis, pulmonary embolism, stroke or other thromboembolic event

OTHER OUTCOMES:
Signs of altered coagulation | 12-24 hours after surgery
  Possible signs hypercoagulopathy in thromboelastometry: EXTEM value of more than 72 mm

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kuitunen, MD, PhD, Study Director — Deputy chief physician
Locations (1):
- Tampere University Hospital, Tampere, Finland